CLINICAL TRIAL: NCT07300241
Title: An Open-Label, First-in-Human, Phase 1/2 Dose Escalation and Expansion Study of NEO-811 in Subjects With Locally Advanced or Metastatic Non-Resectable Clear Cell Renal Cell Carcinoma
Brief Title: Open-Label Phase 1/2 Study of NEO-811 in Subjects With Locally Advanced or Metastatic Non-Resectable Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neomorph, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEO-811-101
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma; RCC; Clear Cell Renal Cell Carcinoma Metastatic; ccRCC; VHL-Associated Clear Cell Renal Cell Carcinoma; VHL-Associated Renal Cell Carcinoma; Kidney Cancer Metastatic; Kidney Cancers
Keywords: ccRCC; Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; VHL; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single agent NEO-811 dose escalation (Experimental): NEO-811
  Interventions: Drug: NEO-811

INTERVENTIONS:
Drug: NEO-811 — NEO-811

SUMMARY:
The NEO-811-101 study is an open-label, first-in-human, Phase 1/2 dose escalation and expansion study of NEO-811 for subjects with locally advanced or metastatic non-resectable clear cell renal cell carcinoma. The study will test NEO-811 initially as a monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with locally advanced or metastatic non-resectable clear cell renal cell carcinoma (ccRCC).
* Subjects must have progressed on or refused standard therapies.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1.
* Estimated life expectancy, in the judgment of the Investigator, of at least 12 weeks.
* Formalin-fixed paraffin-embedded (FFPE) tumor tissue, newly obtained or archival, is mandatory for enrollment to the study.
* Measurable disease as defined by RECIST v1.1.
* Adequate hematologic, hepatic, and renal function defined as:

  * Hemoglobin ≥10 g/dL,
  * Absolute neutrophil count ≥1000 cells/µL,
  * Platelet count ≥100,000/µL,
  * AST and ALT ≤2.5 × ULN, or AST and ALT ≤5 × ULN for subjects with liver metastases,
  * Total bilirubin ≤1.5 × ULN,
  * Estimated glomerular filtration rate (eGFR) ≥60 mL/min.
* Subject can swallow oral medications and does not have a condition that could impair the oral bioavailability of the study drug.
* Other inclusion criteria per protocol.

Exclusion Criteria:

* Non-clear cell predominant RCC histologic subtypes.
* Leptomeningeal disease or symptomatic active CNS metastases with exceptions for asymptomatic treated CNS metastases per protocol.
* Prior or concurrent malignancies with exceptions per protocol.
* History of hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV infection.
* Other exclusion criteria per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs) of NEO-811 as a single agent. | Start of Cycle 1 until at least 30 days following the last dose of the last treatment cycle (each treatment cycle is 21 days).
  TEAEs will be assessed and severity assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 6.0.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of NEO-811 as a single agent. | Start of Cycle 1 until at least 30 days following the last dose of the last treatment cycle (each treatment cycle is 21 days).
  The MTD and/or RP2D of NEO-811 as a single agent will be determined.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of NEO-811. | Start of Cycle 1 until Day 1 of last treatment cycle (each treatment cycle is 21 days).
  Maximum observed plasma concentration (Cmax) of NEO-811 will be determined.
Trough observed plasma concentration (Ctrough) of NEO-811. | Start of Cycle 1 until Day 1 of last treatment cycle (each treatment cycle is 21 days).
  Trough observed plasma concentration (Ctrough) of NEO-811 will be determined.
Time to Cmax (Tmax) of NEO-811. | Start of Cycle 1 until Day 1 of last treatment cycle (each treatment cycle is 21 days).
  Time to Cmax (Tmax) of NEO-811 will be determined.
Area under the concentration time curve (AUC) of NEO-811. | Start of Cycle 1 until Day 1 of last treatment cycle (each treatment cycle is 21 days).
  Area under the concentration time curve (AUC) of NEO-811 will be determined.
Anti-tumor activity of NEO-811 as a single agent. | Start of Cycle 1 until documented disease progression or death, etc. (each treatment cycle is 21 days), estimated as 6-9 months.
  Tumor response will be determined by RECISTv1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Wagner, MD, PhD, Study Director — Neomorph, Inc
Locations (6):
- United States (6):
  - NEO-811 Grand Rapids Site, Grand Rapids, Michigan
  - NEO-811 Long Island Site, Lake Success, New York
  - NEO-811 South Carolina Site, Myrtle Beach, South Carolina
  - NEO-811 Dallas Site, Dallas, Texas
  - NEO-811 Houston Site, Houston, Texas
  - NEO-811 Virginia Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No